CLINICAL TRIAL: NCT00294229
Title: Spinal Manipulative Therapy for Low Back Pain: Randomised Controlled Trial
Brief Title: Spinal Manipulative Therapy for Low Back Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Swiss Society for Manual Therapy (SAMM) (Unknown); Insel Gruppe AG, University Hospital Bern (Other); Wissenschaftlicher Fonds WFR (Unknown)
Responsible Party: Department of Social and Preventive Medicine (ISPM), University of Bern
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEK220_02; INSEL749
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Spinal manipulative therapy; Randomised controlled trial
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: manipulative therapy

SUMMARY:
Context: Acute low back pain (LBP) is a common reason for consultations in primary care. Reducing the pain in the first hours and days and restoring the functional capacity of the lumbar spine may result in a decrease in medical costs and earlier return to work.

Objective: To determine the impact of spinal manipulation on pain and analgesic use in acute low back pain.

DETAILED DESCRIPTION:
Design: Randomised controlled parallel-group trial comparing standard care plus spinal manipulative therapy with standard care alone. Intention-to-treat analysis.

Patients: Outpatients with acute low back pain. Setting: Emergency Department of Bern University Hospital and a primary care practice network.

ELIGIBILITY:
Inclusion criteria:

1. Age between 20 and 55 years
2. Duration of acute low back pain less than 4 weeks
3. Informed consent

Exclusion criteria:

1. Pregnancy
2. Radicular origin of back pain (with irradiation)
3. Cauda equine syndrome
4. Neurologic deficit
5. Epidural glucocorticoid injections in the preceding three months
6. Previous low back surgery
7. Severe osteoporosis
8. Blood-coagulation disorder
9. Allergy to planned rescue medications
10. Suspicion of a specific cause of low back pain (fracture, tumor, infection, inflammatory disease of the spine, HIV-infection) in the patient's history or by physical examination
11. History or signs of severe dysfunction of the liver or kidney

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2003-03; Primary Completion 2006-04 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Back pain overall measured by a numeric rating scale(range 0 to 10)
Analgesic use based on daily equivalence doses (paracetamol, diclofenac and codeine)

SECONDARY OUTCOMES:
Roland Morris Score
Serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Peter M. Villiger, MD, Principal Investigator — Dep. of Rheumatology & Clinical Immunology/Allergology, University Hospital of Berne; Peter Juni, MD, Study Director — Department of Social and Preventive Medicine (ISPM), University of Berne
Locations (1):
- Department of Social and Preventive Medicine (ISPM), University of Bern, Bern, Switzerland